CLINICAL TRIAL: NCT02854371
Title: Evaluation of Hepatic Function Using Gd-EOB-DTPA Enhanced Liver Magnetic Resonance Imaging
Brief Title: Evaluation of Hepatic Function Using Gadoxetic Acid Enhanced MRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-2015-3375
Record Dates: First submitted 2016-07-31; First posted 2016-08-03 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Cirrhosis
Keywords: gadoxetic acid; T1 map; MRI
MeSH Terms: conditions — Fibrosis | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Intervention Model Description: gadoxetic acid MRI and ICG R15 test
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CLD and LC (Experimental): Patients with underlying chronic liver disease. Gadoxetic acid enhanced liver MRI and ICG R15 are performed in this group.
  Interventions: Drug: gadoxetic acid enhanced liver MRI; Drug: ICG R15

INTERVENTIONS:
Drug: gadoxetic acid enhanced liver MRI — Gadoxetic acid enhanced liver MRI is performed and the standard dose of contrast media (0.025mmol/kg) is administered intravenously at a rate of 1mL/sec. Before and after contrast media injection, T1 map sequence is performed to calculate hepatocyte fraction.
  Routine MR sequences (T2WI, T1WI, dual-echo sequence, DWI, MR elastography) are performed according to clinical protocol in the institution.
  Other Names: Primovist; Eovist
Drug: ICG R15 — ICG R15 (Indocyanine green retention test) is performed within 3 days after gadoxetic acid liver MRI, according to clinical standard protocol.
  Other Names: Indocyanine green retention test

SUMMARY:
Liver function is a key factor that can help predict the clinical outcome in patients with cirrhosis. Traditionally, liver function was measured using either indocyanine green (ICG) or other radionucleotides. Recently, gadoxetic acid has been reported to show liver function in several studies. There have been several approaches to measure liver function using gadoxetic acid, and hepatocyte fraction is one of the promising methods. Since gadoxetic acid enhanced liver MRI is clinically used world widely, it would be valuable if we can measure liver function using hepatocyte fraction.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic liver disease or liver cirrhosis
* clinically scheduled for gadoxetic acid enhanced liver MRI
* signed informed consent

Exclusion Criteria:

* under 18 years
* transarterial chemoembolization, radiation therapy for liver or bile duct within 2 weeks
* systemic chemotherapy within 6 weeks
* any contraindication for contrast enhanced MRI
* hepatic iron deposition at prior imaging
* bile duct obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Liver function assessed by hepatocyte fraction | 1 month after MRI
  hepatocyte fraction obtained by T1 map sequence

SECONDARY OUTCOMES:
Liver function assessed by ICG R15 test | 3 days after MRI
Hepatocyte uptake rate | 1 month after MRI
  calculated hepatic uptake rate from T1 map sequence at MRI

OTHER OUTCOMES:
Liver stiffness value (kPa) | 1 month after MRI
  liver stiffness from MR elastography
Spleen stiffness value (kPa) | 1 month after MRI
  spleen stiffness from MR elastography
adverse effect after contrast media administration | within an hour after contrast media administration
adverse effect after ICG administration | within an hour after ICG administration
T2* value (msec) | 1 month after MRI
  T2 star value obtained from Dixon sequence before and after contrast media administration
Bile duct excretion of contrast media on hepatobiliary phase | 1 month after MRI
  five point scale (1: no visualization, 5: opacification of 2nd branch~CBD)
ADC | 1 month after MRI
  apparent diffusion coefficient from DWI sequence using multiple b-values (0~800sec/mm2)
D | 1 month after MRI
  true diffusion coefficient from DWI sequence using multiple b-values (0~800sec/mm2)
D* | 1 month after MRI
  pseudodiffusion coefficient from DWI sequence using multiple b-values (0~800sec/mm2)
f | 1 month after MRI
  perfusion fraction (%) from DWI sequence using multiple b-values (0~800sec/mm2)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No